CLINICAL TRIAL: NCT02298179
Title: A Phase 1 Randomized, Observer Blind, Placebo Controlled, Dosage-Escalation Single Center Study to Evaluate the Safety and Immunogenicity of an RSV Fusion Glycoprotein (F) Subunit Vaccine in Healthy Adults
Brief Title: A Study to Evaluate the Safety and Ability of the Vaccine to Induce Antibodies Against the Respiratory Syncytial Virus in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 205219; 2014-000145-69 (EudraCT Number); V122_01 (Other: Novartis)
Record Dates: First submitted 2014-11-19; First posted 2014-11-21 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Respiratory Syncytial Virus (RSV)
Keywords: Antibodies; Respiratory syncytial virus; Safety; Healthy adults; Immunogenicity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (12):
- RSV F 45 No Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the low dose RSV F subunit vaccine [45 μg], with no adjuvant.
  Interventions: Biological: RSV F subunit 45 μg No adjuvant
- RSV F 45 Alum Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the low dose RSV F subunit vaccine [45 μg], with aluminum hydroxide adjuvant.
  Interventions: Biological: RSV F subunit 45 μg Aluminum hydroxide adjuvant
- RSV F 45 MF59 Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the low dose RSV F subunit vaccine [45 μg], with MF59 adjuvant.
  Interventions: Biological: RSV F subunit 45 μg MF59 adjuvant
- Placebo 1 Group (Placebo Comparator): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of saline solution. Subjects were enrolled in a stepwise dosage escalation manner into one of the three cohorts (Cohort 1: low dosage of RSV F subunit vaccine [45 μg], Cohort 2: middle dosage of RSV F subunit vaccine [90 μg], and Cohort 3: high dosage of RSV F subunit vaccine [135 μg]). This placebo group belongs to Cohort 1.
  Interventions: Drug: Placebo
- RSV F 90 No Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the medium dose RSV F subunit vaccine [90 μg], with no adjuvant.
  Interventions: Biological: RSV F subunit 90 μg No adjuvant
- RSV F 90 Alum Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the medium dose RSV F subunit vaccine [90 μg], with aluminum hydroxide adjuvant.
  Interventions: Biological: RSV F subunit 90 μg Aluminum hydroxide adjuvant
- RSV F 90 MF59 Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the medium dose RSV F subunit vaccine [90 μg], with MF59 adjuvant.
  Interventions: Biological: RSV F subunit 90 μg MF59 adjuvant
- Placebo 2 Group (Placebo Comparator): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of saline solution. Subjects were enrolled in a stepwise dosage escalation manner into one of the three cohorts (Cohort 1: low dosage of RSV F subunit vaccine [45 μg], Cohort 2: middle dosage of RSV F subunit vaccine [90 μg], and Cohort 3: high dosage of RSV F subunit vaccine [135 μg]). This placebo group belongs to Cohort 2.
  Interventions: Drug: Placebo
- RSV F 135 No Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the high dose RSV F subunit vaccine [135 μg], with no adjuvant.
  Interventions: Biological: RSV F subunit 135 μg No adjuvant
- RSV F 135 Alum Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the high dose RSV F subunit vaccine [135 μg], with aluminum hydroxide adjuvant.
  Interventions: Biological: RSV F subunit 135 μg Aluminum hydroxide adjuvant
- RSV F 135 MF59 Adj Group (Experimental): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of the high dose RSV F subunit vaccine [135 μg], with MF59 adjuvant.
  Interventions: Biological: RSV F subunit 135 μg MF59 adjuvant
- Placebo 3 Group (Placebo Comparator): Healthy female and male subjects, 18 to 45 years of age, who received two doses of an intramuscular injection of saline solution. Subjects were enrolled in a stepwise dosage escalation manner into one of the three cohorts (Cohort 1: low dosage of RSV F subunit vaccine [45 μg], Cohort 2: middle dosage of RSV F subunit vaccine [90 μg], and Cohort 3: high dosage of RSV F subunit vaccine [135 μg]). This placebo group belongs to Cohort 3.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: RSV F subunit 45 μg No adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 45 No Adj Group
Biological: RSV F subunit 45 μg Aluminum hydroxide adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 45 Alum Adj Group
Biological: RSV F subunit 45 μg MF59 adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 45 MF59 Adj Group
Biological: RSV F subunit 90 μg No adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 90 No Adj Group
Biological: RSV F subunit 90 μg Aluminum hydroxide adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 90 Alum Adj Group
Biological: RSV F subunit 90 μg MF59 adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 90 MF59 Adj Group
Biological: RSV F subunit 135 μg No adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 135 No Adj Group
Biological: RSV F subunit 135 μg Aluminum hydroxide adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 135 Alum Adj Group
Biological: RSV F subunit 135 μg MF59 adjuvant — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Arms: RSV F 135 MF59 Adj Group
Drug: Placebo — 2 doses of 0.5 milliliters (mL) each of injectable solution administered intramuscularly, in the deltoid muscle, preferably in the non-dominant arm.
  Other Names: Sterile saline 0.9%
  Arms: Placebo 1 Group; Placebo 2 Group; Placebo 3 Group

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of two doses of the investigational RSV F subunit vaccine administered intramuscularly (IM). In this current Phase 1, first-in-human study, the three different antigen amounts that have been selected will be evaluated in a stepwise manner in three different cohorts (Cohort 1: low dosage of RSV F subunit vaccine, Cohort 2: middle dosage of RSV F subunit vaccine, and Cohort 3: high dosage of RSV F subunit vaccine). In addition, the effect of an adjuvant, either aluminum hydroxide or MF59, and antibody kinetics post-vaccination at different time points will be evaluated as compared to unadjuvanted RSV F subunit vaccine at the same dosage levels.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males and non-pregnant females 18 to 45 years of age at time of enrollment.
2. Individuals who have given written consent after the nature of the study has been explained according to local regulatory requirements.
3. Individuals in good health as determined by the outcome of the medical history, physical examination and clinical judgment of the investigator.
4. Individuals who can comply with the study procedures and are available for follow up.

Exclusion Criteria:

1. Individuals with any severe chronic or acute disease.
2. Individuals with a history of illness or with an ongoing illness that may pose additional risk to the subject if he/she participates in the study, including the following:

   * History of any chronic respiratory illness, including current diagnosis of asthma within 2 years, exercise induced wheezing, reactive airway disease, emphysema, chronic bronchitis, cystic fibrosis or chronic obstructive pulmonary disease (COPD).
   * Any respiratory illness within 7 days prior to receiving the first study injection.
   * Any active pulmonary infection or other inflammatory conditions, even in the absence of febrile episodes, within 14 days prior to the first study injection.
   * Hepatitis B or hepatitis C infection.
3. Individuals who have had a malignancy or lymphoproliferative disorder within the past 5 years.
4. Individuals with known or suspected impairment of the immune system including but not limited to HIV, autoimmune disorders, immunosuppressive therapy, and diabetes mellitus.
5. Individuals with any history of progressive or severe neurologic disorder, seizure disorder or Guillian-Barré syndrome.
6. Individuals with a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
7. Individuals with a BMI > 35 kg/m2. BMI is to be calculated by the following formula: subject weight at baseline divided by subject height in meters multiplied by the subject height in meters. The numerical result will be rounded to the nearest 0.1.
8. Individuals who are allergic to any of the vaccine components, or with a history of anaphylaxis after vaccination.
9. Individuals who during the 90 days prior to enrollment receive any medications or other treatments that may adversely affect the immune system such as allergy injections, immune globulin, interferon, immunomodulators, cytotoxic drugs or other drugs known to be frequently associated with significant major organ toxicity.
10. Individuals who receive systemic immunosuppressive agents including steroids. Prior corticosteroid therapy should be discontinued 28 days prior to enrollment. Individuals using inhaled or topical corticosteroids will be permitted.
11. Receipt or donation of blood or blood products 8 weeks prior to vaccination or planned receipt or donation during the study period.
12. Individuals participating in any clinical trial with another investigational product 28 days prior to receiving the first study vaccination or intent to participate in another clinical study at any time during the conduct of this study.
13. Individuals who have received any vaccine 28 days prior to enrollment in this study, or who plan to receive any non-study vaccines within 28 days of the second dose of study vaccine.
14. Individuals with any clinically significant abnormal safety laboratory result, as judged by the investigator.
15. If female, 'of childbearing potential', sexually active and has not used any of the 'acceptable contraceptive methods' for at least two months prior to study entry.

    Childbearing potential is defined as status post onset of menarche and not meeting any of the following conditions: menopausal for at least two years; sterile status after bilateral tubal ligation for at least one year, immediately after bilateral oophorectomy or after hysterectomy.

    Acceptable methods of birth control are defined as one or more of the following:
    * Hormonal contraceptives.
    * Barrier each and every time during intercourse.
    * Intrauterine device (IUD).
    * Monogamous relationship with vasectomized partner. Partner must have been vasectomized for at least six months prior to subject's study entry.
16. If female subject of childbearing potential and have a positive urine pregnancy test prior to study vaccinations, or are currently lactating.
17. If female of childbearing potential and sexually active, refusal to use an 'acceptable contraceptive method' through to three weeks after last study vaccination.
18. Individuals with behavioral or cognitive impairment or psychiatric disease that, in the opinion of the investigator, may interfere with the subject's ability to participate in the study.
19. Individuals with a history of drug or alcohol abuse within the past 2 years.
20. Individuals who are acting as study personnel or immediate family members or the spouse of study personnel.
21. Individuals with a body temperature ≥38 °C (≥100.4◦F) within 3 days of intended study vaccination.
22. Individuals with any condition that, in the opinion of the investigator, would interfere with the primary study objectives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2014-12-19 (Actual); Primary Completion 2017-03-27 (Actual); Study Completion 2017-03-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Ghent, Belgium

REFERENCES:
- [Derived] Schneikart G, Tavarini S, Sammicheli C, Torricelli G, Guidotti S, Andreano E, Buricchi F, D'Oro U, Finco O, Bardelli M. The respiratory syncytial virus fusion protein-specific B cell receptor repertoire reshaped by post-fusion subunit vaccination. Vaccine. 2020 Nov 25;38(50):7916-7927. doi: 10.1016/j.vaccine.2020.10.062. Epub 2020 Oct 29. PMID 33131932
- [Derived] Leroux-Roels G, De Boever F, Maes C, Nguyen TL, Baker S, Gonzalez Lopez A. Safety and immunogenicity of a respiratory syncytial virus fusion glycoprotein F subunit vaccine in healthy adults: Results of a phase 1, randomized, observer-blind, controlled, dosage-escalation study. Vaccine. 2019 May 6;37(20):2694-2703. doi: 10.1016/j.vaccine.2019.04.011. Epub 2019 Apr 12. PMID 30987852

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from one site in Belgium.
Pre-assignment Details: All subjects enrolled were included in the trial.
Period: Overall Study
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Started | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Completed | 24 | 24 | 23 | 24 | 24 | 24 | 24 | 23 | 24 | 24 | 24 | 24
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group | Total
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 288
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.6 (6.8) | 27.7 (6.55) | 30.2 (7.9) | 30.3 (7.62) | 30.4 (8.31) | 31.2 (7.47) | 27.6 (6.84) | 28 (7.3) | 28.3 (6.8) | 29.5 (6.98) | 32.9 (8.46) | 27.9 (5.86) | 29.13 (7.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 18 | 18 | 16 | 18 | 15 | 14 | 22 | 18 | 20 | 20 | 216
  Male | 4 | 7 | 6 | 6 | 8 | 6 | 9 | 10 | 2 | 6 | 4 | 4 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  BLACK OR AFRICAN AMERICAN | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  WHITE | 23 | 22 | 24 | 24 | 24 | 24 | 24 | 23 | 24 | 24 | 24 | 24 | 284
  NOT SPECIFIED | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of the Serum Anti-RSV Neutralizing Antibody (NAb) Titers
Description: Immunogenicity was measured in terms of the Geometric mean titers (GMTs) of the serum anti-RSV neutralizing antibody (NAb) titers at Day 57 (28 days after the second dose).
Time Frame: At Day 57
Population: The analysis was based on the Per-Protocol Set (PPS), which included all subjects in the Full Analysis Set (FAS) Immunogenicity population who were not excluded due to the reasons defined prior to unblinding or analysis and for whom immunogenicity data were available at Day 57.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
Titers | 864 [692 to 1077] | 914 [738 to 1134] | 843 [673 to 1057] | 234 [169 to 324] | 844 [665 to 1072] | 746 [587 to 947] | 944 [735 to 1213] | 253 [189 to 337] | 903 [729 to 1119] | 1212 [974 to 1509] | 1316 [1066 to 1623] | 254 [183 to 354]

2. Primary Outcome: Percentage of Subjects With a ≥ 4-fold Increase in Serum Anti-RSV NAb Titers
Description: Immunogenicity was measured in terms of percentage of subjects with a ≥ 4-fold increase in serum anti-RSV NAb titers, from Day 1 (baseline) to Day 57 (28 days after the second dose).
Time Frame: At Day 57
Population: The analysis was based on PPS, which included all subjects in the FAS Immunogenicity population who were not excluded due to reasons defined prior to unblinding or analysis and and for whom immunogenicity results collected from Day 1 (baseline) up to Day 57 were available at Day 1 and Day 57.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
Percentage of subjects | 45 [24.4 to 67.8] | 54 [32.8 to 74.4] | 36 [17.2 to 59.3] | 0 [0.0 to 14.8] | 25 [9.8 to 46.7] | 29 [12.6 to 51.1] | 41 [20.7 to 63.6] | 0 [0.0 to 14.8] | 17 [5.0 to 38.8] | 45 [24.4 to 67.8] | 46 [25.6 to 67.2] | 0 [0.0 to 14.2]

3. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: Assessed solicited local symptoms were: induration, swelling, erythema and pain. Any induration/swelling/erythema = induration/swelling/erythema spreading beyond 25 millimeters (mm) of injection site. Any pain = occurrence of the symptom regardless of intensity grade.
Time Frame: Within 30 minutes after each vaccination
Population: The analysis was based on the Solicited Safety set, which included all subjects in the Exposed population who provided post-vaccination reactogenicity data after each vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Induration (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain (1st) | 3 | 1 | 0 | 3 | 1 | 4 | 4 | 2 | 2 | 2 | 1 | 3
  Any Induration (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Induration (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Swelling (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Erythema (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Pain (2nd) | 2 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 0 | 2

4. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: as for outcome 3
Time Frame: From Day 1 (6 hour) through Day 3 after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Induration (1st) | 0 | 3 | 2 | 0 | 1 | 2 | 3 | 0 | 0 | 2 | 2 | 1
  Any Swelling (1st) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
  Any Erythema (1st) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
  Any Pain (1st) | 12 | 21 | 19 | 2 | 10 | 18 | 20 | 2 | 12 | 22 | 18 | 5
  Any Induration (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Induration (2nd) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1
  Any Swelling (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Swelling (2nd) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Any Erythema (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Erythema (2nd) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Any Pain (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Pain (2nd) | 13 | 11 | 13 | 4 | 16 | 12 | 13 | 0 | 15 | 11 | 14 | 5

5. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: as for outcome 3
Time Frame: From Day 4 through Day 7 after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Induration (1st) | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any Swelling (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
  Any Erythema (1st) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any Pain (1st) | 8 | 7 | 4 | 0 | 7 | 8 | 3 | 0 | 9 | 5 | 4 | 0
  Any Induration (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Induration (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Swelling (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Swelling (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Erythema (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Pain (2nd) | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1

6. Primary Outcome: Number of Subjects With Any Solicited Local Symptoms
Description: as for outcome 3
Time Frame: From Day 1 (6 hours) to Day 7 after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Induration (1st) | 0 | 4 | 2 | 0 | 1 | 2 | 3 | 0 | 0 | 2 | 2 | 1
  Any Swelling (1st) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 1 | 0
  Any Erythema (1st) | 1 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 0 | 0
  Any Pain (1st) | 14 | 21 | 19 | 2 | 11 | 18 | 20 | 2 | 13 | 22 | 18 | 5
  Any Induration (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Induration (2nd) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 1 | 1
  Any Swelling (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Swelling (2nd) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
  Any Erythema (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Erythema (2nd) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Any Pain (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Pain (2nd) | 13 | 11 | 13 | 4 | 16 | 12 | 13 | 0 | 15 | 11 | 14 | 5

7. Primary Outcome: Number of Subjects With Any Solicited Systemic Symptoms and Other Indicators of Reactogenicity
Description: Assessed solicited systemic symptoms were: nausea, fatigue, myalgia, arthralgia, headache, fever (body temperature ≥ 38.0°C), chills, coughing, diarrhea, rhinorrhea and wheezing. Other solicited data included: prevention of pain and/or fever and treatment of pain and/or fever. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: Within 30 minutes after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Nausea (1st) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Any Fatigue (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache (1st) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fever (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Coughing (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Diarrhea (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Rhinorrhea (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Wheezing (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (1st) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Nausea (2nd) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Fatigue (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Myalgia (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Arthralgia (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Headache (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Fever (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Fever (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Chills (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Coughing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Coughing (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Diarrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Diarrhea (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Rhinorrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Rhinorrhea (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Wheezing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Any Wheezing (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Pain/Fever prevention (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 23 | 24
  Pain/Fever treatment (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Primary Outcome: Number of Subjects With Any Solicited Systemic Symptoms and Other Indicators of Reactogenicity
Description: as for outcome 7
Time Frame: From Day 1 (6 hours) through Day 3 after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Nausea (1st) | 1 | 1 | 3 | 2 | 4 | 0 | 1 | 1 | 1 | 3 | 4 | 2
  Any Fatigue (1st) | 6 | 7 | 8 | 8 | 7 | 7 | 9 | 7 | 4 | 7 | 7 | 5
  Any Myalgia (1st) | 1 | 1 | 4 | 0 | 1 | 3 | 3 | 0 | 2 | 5 | 4 | 0
  Any Arthralgia (1st) | 3 | 0 | 4 | 0 | 2 | 2 | 1 | 0 | 1 | 1 | 3 | 1
  Any Headache (1st) | 6 | 5 | 1 | 5 | 5 | 6 | 7 | 5 | 4 | 7 | 9 | 2
  Any Fever (1st) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills (1st) | 2 | 1 | 5 | 0 | 2 | 1 | 0 | 1 | 2 | 3 | 3 | 0
  Any Coughing (1st) | 5 | 3 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 4 | 4 | 4
  Any Diarrhea (1st) | 4 | 0 | 0 | 3 | 4 | 2 | 2 | 1 | 0 | 4 | 3 | 0
  Any Rhinorrhea (1st) | 7 | 5 | 4 | 4 | 5 | 3 | 4 | 6 | 3 | 8 | 6 | 4
  Any Wheezing (1st) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Pain/Fever prevention (1st) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (1st) | 3 | 0 | 0 | 0 | 4 | 1 | 2 | 0 | 1 | 2 | 3 | 1
  Any Nausea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Nausea (2nd) | 1 | 1 | 1 | 2 | 2 | 3 | 1 | 4 | 1 | 2 | 1 | 2
  Any Fatigue (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Fatigue (2nd) | 3 | 4 | 6 | 6 | 7 | 4 | 1 | 6 | 3 | 3 | 6 | 5
  Any Myalgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Myalgia (2nd) | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 1 | 1 | 0 | 2 | 1
  Any Arthralgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Arthralgia (2nd) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0
  Any Headache (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Headache (2nd) | 3 | 4 | 6 | 4 | 6 | 5 | 0 | 5 | 3 | 4 | 4 | 1
  Any Fever (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Fever (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any Chills (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Chills (2nd) | 1 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 2
  Any Coughing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Coughing (2nd) | 2 | 3 | 3 | 2 | 2 | 1 | 1 | 1 | 2 | 1 | 3 | 1
  Any Diarrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Diarrhea (2nd) | 1 | 1 | 0 | 3 | 1 | 1 | 0 | 3 | 0 | 2 | 1 | 2
  Any Rhinorrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Rhinorrhea (2nd) | 6 | 8 | 3 | 3 | 3 | 2 | 3 | 1 | 2 | 3 | 5 | 4
  Any Wheezing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Wheezing (2nd) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention (2nd): number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24 | 22 | 23 | 24 | 23 | 24 | 24
  Pain/Fever prevention (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (2nd): number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24 | 22 | 23 | 24 | 23 | 24 | 24
  Pain/Fever treatment (2nd) | 2 | 3 | 2 | 3 | 1 | 3 | 0 | 0 | 2 | 3 | 1 | 1

9. Primary Outcome: Number of Subjects With Any Solicited Systemic Symptoms and Other Indicators of Reactogenicity
Description: as for outcome 7
Time Frame: From Day 4 through Day 7 after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Nausea (1st): number analyzed (Participants) | 24 | 24 | 23 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
  Any Nausea (1st) | 1 | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 1 | 2 | 3 | 3
  Any Fatigue (1st) | 2 | 3 | 6 | 8 | 4 | 5 | 7 | 7 | 4 | 4 | 5 | 4
  Any Myalgia (1st) | 1 | 0 | 1 | 2 | 1 | 2 | 2 | 1 | 1 | 0 | 2 | 1
  Any Arthralgia (1st) | 2 | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 1
  Any Headache (1st) | 3 | 1 | 1 | 7 | 4 | 6 | 7 | 7 | 2 | 4 | 4 | 3
  Any Fever (1st) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Any Chills (1st) | 1 | 0 | 2 | 0 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 1
  Any Coughing (1st) | 7 | 3 | 6 | 1 | 3 | 4 | 4 | 1 | 3 | 7 | 5 | 6
  Any Diarrhea (1st) | 2 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 1 | 1 | 2 | 0
  Any Rhinorrhea (1st) | 7 | 6 | 8 | 6 | 4 | 6 | 6 | 6 | 3 | 7 | 9 | 6
  Any Wheezing (1st) | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0 | 1
  Pain/Fever prevention (1st) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (1st) | 1 | 0 | 0 | 0 | 2 | 2 | 2 | 0 | 1 | 0 | 1 | 1
  Any Nausea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Nausea (2nd) | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 5 | 4 | 2 | 2 | 3
  Any Fatigue (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Fatigue (2nd) | 5 | 3 | 2 | 3 | 5 | 2 | 1 | 3 | 2 | 2 | 5 | 3
  Any Myalgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Myalgia (2nd) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 1
  Any Arthralgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Arthralgia (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1
  Any Headache (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Headache (2nd) | 2 | 5 | 0 | 4 | 5 | 2 | 3 | 2 | 3 | 3 | 3 | 4
  Any Fever (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Fever (2nd) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Any Chills (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Chills (2nd) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1
  Any Coughing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Coughing (2nd) | 3 | 2 | 3 | 3 | 3 | 1 | 0 | 0 | 1 | 4 | 1 | 2
  Any Diarrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Diarrhea (2nd) | 1 | 0 | 0 | 2 | 1 | 0 | 1 | 3 | 0 | 2 | 2 | 1
  Any Rhinorrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Rhinorrhea (2nd) | 7 | 4 | 3 | 5 | 5 | 4 | 3 | 2 | 3 | 5 | 2 | 4
  Any Wheezing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Wheezing (2nd) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Pain/Fever prevention (2nd): number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24 | 22 | 23 | 24 | 23 | 24 | 24
  Pain/Fever prevention (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (2nd): number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24 | 22 | 23 | 24 | 23 | 24 | 24
  Pain/Fever treatment (2nd) | 0 | 1 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 3

10. Primary Outcome: Number of Subjects With Any Solicited Systemic Symptoms and Other Indicators of Reactogenicity
Description: as for outcome 7
Time Frame: From Day 1 (6 hours) to Day 7 after each vaccination
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any Nausea (1st) | 2 | 1 | 3 | 3 | 5 | 2 | 3 | 3 | 2 | 4 | 5 | 3
  Any Fatigue (1st) | 7 | 8 | 10 | 10 | 9 | 10 | 10 | 8 | 5 | 7 | 9 | 7
  Any Myalgia (1st) | 1 | 1 | 5 | 2 | 2 | 5 | 4 | 1 | 3 | 5 | 4 | 1
  Any Arthralgia (1st) | 3 | 0 | 4 | 1 | 3 | 2 | 2 | 0 | 1 | 2 | 4 | 2
  Any Headache (1st) | 7 | 5 | 2 | 11 | 8 | 9 | 10 | 9 | 5 | 9 | 10 | 5
  Any Fever (1st) | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 1
  Any Chills (1st) | 2 | 1 | 5 | 0 | 3 | 2 | 2 | 1 | 2 | 4 | 4 | 1
  Any Coughing (1st) | 8 | 5 | 6 | 2 | 3 | 5 | 4 | 1 | 3 | 7 | 6 | 6
  Any Diarrhea (1st) | 4 | 0 | 0 | 3 | 5 | 2 | 2 | 2 | 1 | 4 | 4 | 0
  Any Rhinorrhea (1st) | 8 | 9 | 9 | 7 | 7 | 7 | 7 | 10 | 4 | 9 | 10 | 6
  Any Wheezing (1st) | 2 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 1 | 1
  Pain/Fever prevention (1st) | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (1st) | 3 | 0 | 0 | 0 | 5 | 2 | 4 | 0 | 2 | 2 | 3 | 2
  Any Nausea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Nausea (2nd) | 1 | 2 | 1 | 2 | 2 | 3 | 1 | 6 | 5 | 4 | 3 | 3
  Any Fatigue (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Fatigue (2nd) | 6 | 5 | 7 | 7 | 8 | 4 | 2 | 6 | 4 | 4 | 8 | 6
  Any Myalgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Myalgia (2nd) | 1 | 0 | 1 | 3 | 1 | 1 | 0 | 2 | 2 | 1 | 2 | 1
  Any Arthralgia (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Arthralgia (2nd) | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 1 | 2 | 2 | 1
  Any Headache (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Headache (2nd) | 4 | 7 | 6 | 6 | 9 | 5 | 3 | 6 | 5 | 7 | 6 | 4
  Any Fever (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Fever (2nd) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Any Chills (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Chills (2nd) | 2 | 0 | 1 | 2 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 2
  Any Coughing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Coughing (2nd) | 3 | 3 | 4 | 4 | 4 | 2 | 1 | 1 | 2 | 4 | 3 | 2
  Any Diarrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Diarrhea (2nd) | 2 | 1 | 0 | 3 | 1 | 1 | 1 | 3 | 0 | 3 | 2 | 3
  Any Rhinorrhea (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Rhinorrhea (2nd) | 7 | 8 | 4 | 5 | 6 | 5 | 3 | 2 | 4 | 6 | 6 | 6
  Any Wheezing (2nd): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any Wheezing (2nd) | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Pain/Fever prevention (2nd): number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24 | 22 | 23 | 24 | 23 | 24 | 24
  Pain/Fever prevention (2nd) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment (2nd): number analyzed (Participants) | 23 | 23 | 23 | 24 | 24 | 24 | 22 | 23 | 24 | 23 | 24 | 24
  Pain/Fever treatment (2nd) | 2 | 3 | 2 | 4 | 2 | 3 | 1 | 1 | 2 | 3 | 1 | 3

11. Primary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
  Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: From Day 1 to Day 28 after each vaccination
Population: The analysis was based on the Unsolicited Safety Set, which included all subjects in the Exposed population with unsolicited AE data collected after each vaccination.
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any AE(s) (1st vacc.) | 17 | 15 | 14 | 17 | 15 | 14 | 16 | 14 | 13 | 14 | 15 | 17
  Any AE(s) (2nd vacc.): number analyzed (Participants) | 23 | 24 | 23 | 24 | 24 | 24 | 22 | 24 | 24 | 23 | 24 | 24
  Any AE(s) (2nd vacc.) | 8 | 12 | 16 | 13 | 13 | 7 | 6 | 13 | 10 | 9 | 13 | 10

12. Primary Outcome: Number of Subjects With Serious Adverse Events (SAEs) and Other Significant AE(s)
Description: SAEs assessed include medical occurrences that resulted in death, were life-threatening, required hospitalization or prolongation of hospitalization or resulted in disability/incapacity, congenital anomaly or birth defect. Any SAE = occurrence of the SAE regardless of intensity grade. Possibly or probably related SAE = SAE assessed by the investigator as possibly or probably related to the study vaccination.
  Other significant AE(s) assessed include unsolicited medically attended AEs, unsolicited AEs leading to study withdrawal, new onset of chronic diseases (NOCDs) and adverse events of special interest (AESIs). Medically attended AE = an adverse event that leads to an unscheduled visit to a healthcare practitioner. NOCD = an adverse event that represents a new diagnosis of a chronic medical condition that was not present or suspected in a subject prior to study enrollment.
Time Frame: From study start (Day 1) until study completion (Day 394)
Population: The analysis was based on the Unsolicited Safety Set, which included all subjects in the Exposed population with unsolicited AE data collected from study start (Day 1) until study completion (Day 394).
Measure: Count of Participants; unit: Participants
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24 | 24
Participants
  Any SAE(s) | 1 | 1 | 1 | 0 | 1 | 0 | 4 | 0 | 1 | 2 | 0 | 0
  Possibly/probably related SAE(s) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Any medically attended AE(s) | 10 | 11 | 12 | 17 | 17 | 9 | 16 | 15 | 15 | 15 | 12 | 11
  Any AE(s) leading to study withdrawal | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Any NOCD(s) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Any AESI(s) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Geometric Mean Titers (GMTs) of the Serum Anti-RSV Neutralizing Antibody (NAb) Titers
Description: Immunogenicity was measured in terms of GMTs of the serum anti-RSV neutralizing antibody (NAb) titers at Day 1, Day 29 (28 days after the first dose) and Day 181 (six months after the first dose).
Time Frame: At Day 1, Day 29 and Day 181
Population: The analysis was based on the PPS, which included all subjects in the FAS Immunogenicity population who were not excluded due to reasons defined prior to unblinding or analysis and for whom immunogenicity data were available at Day 1, Day 29 and at Day 181.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Titers
  Anti-RSV NAb, Day 1 | 237 [162 to 345] | 184 [127 to 266] | 340 [233 to 497] | 215 [155 to 298] | 289 [209 to 399] | 280 [203 to 387] | 254 [181 to 356] | 233 [175 to 308] | 338 [240 to 476] | 332 [236 to 467] | 380 [272 to 531] | 292 [217 to 392]
  Anti-RSV NAb, Day 29 | 893 [702 to 1136] | 947 [745 to 1203] | 983 [769 to 1257] | 236 [171 to 326] | 1110 [869 to 1419] | 981 [768 to 1253] | 1208 [935 to 1561] | 242 [188 to 313] | 1123 [872 to 1447] | 1602 [1243 to 2064] | 1551 [1210 to 1988] | 286 [218 to 374]
  Anti-RSV NAb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  Anti-RSV NAb, Day 181 | 576 [463 to 717] | 587 [474 to 726] | 450 [360 to 563] | 234 [166 to 328] | 684 [558 to 840] | 627 [508 to 774] | 597 [478 to 745] | 260 [202 to 335] | 687 [566 to 834] | 788 [649 to 957] | 764 [632 to 923] | 248 [191 to 321]

14. Secondary Outcome: Percentage of Subjects With a ≥ 4-fold Increase in Serum Anti-RSV NAb Titer
Description: Immunogenicity was measured in terms of percentage of subjects with a ≥ 4-fold increase in serum anti-RSV NAb titers from Day 1 to Day 29 (28 days after the first dose) and from Day 1 to Day 181 (six months after the first dose).
Time Frame: At Day 29 and at Day 181
Population: The analysis was based on the PPS, which included all subjects in the FAS Immunogenicity population who were not excluded due to reasons defined prior to unblinding or analysis and for whom immunogenicity data were available at Day 1, Day 29 and Day 181.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Percentage of subjects
  Anti-RSV NAb, Day 29 | 48 [26.8 to 69.4] | 58 [36.6 to 77.9] | 30 [13.2 to 52.9] | 0 [0.0 to 14.8] | 25 [9.8 to 46.7] | 42 [22.1 to 63.4] | 50 [28.2 to 71.8] | 0 [0.0 to 14.2] | 35 [16.4 to 57.3] | 57 [34.5 to 76.8] | 42 [22.1 to 63.4] | 0 [0.0 to 14.2]
  Anti-RSV NAb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  Anti-RSV NAb, Day 181 | 32 [13.9 to 54.9] | 29 [12.6 to 51.1] | 5 [0.12 to 22.8] | 0 [0.0 to 15.4] | 17 [5.0 to 38.8] | 14 [2.9 to 34.9] | 15 [3.2 to 37.9] | 0 [0.0 to 14.8] | 14 [2.9 to 34.9] | 27 [10.7 to 50.2] | 17 [5.0 to 38.8] | 0 [0.0 to 14.2]

15. Secondary Outcome: Percentage of Subjects With Serum Anti-RSV NAb Titers Greater Than the 3rd Quartile of Serum Anti-RSV NAb Titers at Day 1
Description: Immunogenicity was measured in terms of the percentage of subjects at Day 29 (28 days after the first dose), Day 57 (28 days after the second dose) and Day 181 (six months after the first dose) with serum anti-RSV NAb titers greater than the 3rd quartile of serum anti-RSV NAb titers at Day 1 (baseline).
Time Frame: At Day 29, Day 57 and Day 181
Population: The analysis was based on the PPS, which included all subjects in the FAS Immunogenicity population who were not excluded due to reasons defined prior to unblinding or analysis and for whom immunogenicity data were available at Day 1, Day 29, Day 57 and Day 181.
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Percentage of subjects
  Anti-RSV NAb, Day 29 | 78 [56.3 to 92.5] | 83 [62.6 to 95.3] | 100 [85.2 to 100.0] | 17 [5.0 to 38.8] | 92 [73.0 to 99.0] | 92 [73.0 to 99.0] | 91 [70.8 to 98.9] | 13 [2.7 to 32.4] | 91 [72.0 to 98.9] | 100 [85.2 to 100.0] | 100 [85.8 to 100.0] | 25 [9.8 to 46.7]
  Anti-RSV NAb, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  Anti-RSV NAb, Day 57 | 95 [77.2 to 99.88] | 79 [57.8 to 92.9] | 95 [77.2 to 99.88] | 9 [1.1 to 28.0] | 83 [62.6 to 95.3] | 79 [57.8 to 92.9] | 95 [77.2 to 99.88] | 17 [5.0 to 38.8] | 91 [72.0 to 98.9] | 91 [70.8 to 98.9] | 100 [85.8 to 100.0] | 25 [9.8 to 46.7]
  Anti-RSV NAb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  Anti-RSV NAb, Day 181 | 64 [40.7 to 82.8] | 50 [29.1 to 70.9] | 64 [40.7 to 82.8] | 18 [5.2 to 40.3] | 87 [66.4 to 97.2] | 73 [49.8 to 89.3] | 65 [40.8 to 84.6] | 13 [2.8 to 33.6] | 68 [45.1 to 86.1] | 82 [59.7 to 94.8] | 74 [51.6 to 89.8] | 17 [4.7 to 37.4]

16. Secondary Outcome: Geometric Mean Titers (GMTs) of the Serum Total Binding Antibody to Each of the RSV Proteins F, G and N
Description: Immunogenicity was measured in terms of the geometric mean titers (GMTs) of the serum total binding antibody to each of the RSV proteins F, G and N at Day 1 (baseline), Day 29 (28 days after the first dose), Day 57 (28 days after the second dose) and Day 181 (six months after the first dose).
Time Frame: At Day 1, Day 29, Day 57 and Day 181
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Titers
  RSV Protein F, Day 1 | 671 [470 to 958] | 838 [591 to 1188] | 916 [642 to 1309] | 714 [530 to 961] | 697 [483 to 1005] | 730 [506 to 1053] | 751 [512 to 1101] | 727 [574 to 921] | 880 [639 to 1210] | 685 [498 to 942] | 910 [666 to 1244] | 750 [586 to 959]
  RSV Protein F, Day 29 | 9641 [7964 to 11671] | 11131 [9244 to 13403] | 11639 [9620 to 14080] | 675 [504 to 905] | 13017 [11147 to 15201] | 10694 [9158 to 12488] | 12841 [10921 to 15099] | 684 [515 to 909] | 13252 [11607 to 15130] | 13514 [11824 to 15446] | 13541 [11890 to 15421] | 851 [617 to 1174]
  RSV Protein F, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein F, Day 57 | 8064 [6645 to 9786] | 9707 [8073 to 11672] | 10182 [8395 to 12349] | 757 [541 to 1060] | 11470 [9660 to 13618] | 10131 [8533 to 12028] | 11588 [9686 to 13864] | 660 [505 to 864] | 11302 [10022 to 12746] | 13483 [11909 to 15264] | 12158 [10806 to 13680] | 791 [596 to 1050]
  RSV Protein F, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein F, Day 181 | 4904 [3848 to 6250] | 6584 [5226 to 8294] | 5312 [4171 to 6765] | 690 [506 to 942] | 6908 [5627 to 8480] | 6271 [5087 to 7730] | 5824 [4675 to 7256] | 763 [596 to 978] | 6157 [5018 to 7556] | 8651 [7038 to 10635] | 7041 [5765 to 8599] | 833 [663 to 1046]
  RSV Protein Ga, Day 1 | 64 [42 to 97] | 57 [38 to 85] | 60 [40 to 91] | 44 [29 to 68] | 53 [36 to 78] | 55 [38 to 81] | 48 [32 to 72] | 57 [39 to 84] | 55 [38 to 79] | 51 [35 to 73] | 65 [46 to 93] | 49 [31 to 79]
  RSV Protein Ga, Day 29 | 64 [56 to 73] | 55 [49 to 62] | 59 [52 to 66] | 43 [27 to 67] | 50 [43 to 59] | 47 [41 to 55] | 46 [39 to 53] | 51 [34 to 75] | 59 [51 to 69] | 47 [41 to 54] | 57 [50 to 66] | 55 [34 to 89]
  RSV Protein Ga, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Ga, Day 57 | 62 [53 to 71] | 53 [47 to 61] | 55 [48 to 64] | 42 [28 to 65] | 49 [43 to 56] | 46 [40 to 53] | 44 [38 to 51] | 46 [31 to 68] | 60 [51 to 71] | 43 [36 to 50] | 51 [43 to 59] | 52 [32 to 83]
  RSV Protein Ga, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Ga, Day 181 | 61 [51 to 73] | 55 [46 to 65] | 58 [49 to 69] | 40 [26 to 60] | 49 [40 to 59] | 54 [44 to 66] | 47 [39 to 58] | 60 [44 to 82] | 54 [43 to 67] | 45 [36 to 56] | 53 [43 to 66] | 49 [31 to 76]
  RSV Protein Gb, Day 1 | 109 [72 to 166] | 105 [70 to 159] | 120 [79 to 183] | 99 [70 to 139] | 107 [72 to 159] | 97 [65 to 145] | 123 [81 to 187] | 100 [67 to 151] | 104 [68 to 161] | 91 [59 to 139] | 112 [73 to 170] | 80 [49 to 129]
  RSV Protein Gb, Day 29 | 122 [107 to 139] | 96 [84 to 109] | 112 [98 to 127] | 102 [70 to 147] | 95 [82 to 110] | 92 [79 to 107] | 87 [74 to 102] | 90 [58 to 140] | 107 [91 to 127] | 97 [82 to 114] | 109 [93 to 129] | 91 [54 to 153]
  RSV Protein Gb, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Gb, Day 57 | 123 [105 to 144] | 97 [83 to 113] | 106 [91 to 124] | 109 [76 to 157] | 93 [82 to 105] | 89 [79 to 101] | 89 [78 to 101] | 78 [49 to 125] | 106 [93 to 121] | 87 [76 to 99] | 89 [78 to 102] | 87 [54 to 140]
  RSV Protein Gb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Gb, Day 181 | 106 [87 to 128] | 94 [78 to 112] | 101 [84 to 122] | 98 [70 to 139] | 99 [85 to 116] | 112 [95 to 131] | 93 [79 to 111] | 101 [72 to 141] | 102 [88 to 119] | 94 [80 to 109] | 98 [84 to 113] | 87 [53 to 141]
  RSV Protein N, Day 1 | 480 [338 to 682] | 525 [373 to 741] | 586 [413 to 832] | 444 [357 to 554] | 418 [308 to 569] | 486 [358 to 661] | 508 [368 to 700] | 424 [305 to 590] | 462 [352 to 606] | 417 [318 to 547] | 569 [437 to 742] | 392 [299 to 513]
  RSV Protein N, Day 29 | 592 [523 to 670] | 434 [385 to 490] | 467 [412 to 529] | 418 [325 to 537] | 439 [378 to 509] | 470 [405 to 546] | 443 [379 to 518] | 412 [299 to 568] | 524 [458 to 600] | 417 [364 to 478] | 471 [412 to 539] | 456 [336 to 619]
  RSV Protein N, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein N, Day 57 | 580 [498 to 676] | 461 [398 to 534] | 513 [440 to 599] | 457 [351 to 596] | 396 [348 to 449] | 423 [373 to 480] | 401 [351 to 458] | 345 [255 to 465] | 514 [459 to 576] | 426 [379 to 479] | 439 [392 to 490] | 418 [319 to 549]
  RSV Protein N, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein N, Day 181 | 524 [448 to 613] | 391 [336 to 454] | 420 [359 to 491] | 421 [337 to 528] | 397 [343 to 460] | 484 [416 to 562] | 425 [363 to 497] | 454 [340 to 608] | 493 [435 to 558] | 454 [400 to 514] | 458 [405 to 518] | 439 [338 to 571]

17. Secondary Outcome: Percentage of Subjects With a ≥ 4-fold Increase in Serum Total Binding Antibody to Each of the RSV Proteins F, G and N
Description: Immunogenicity was measured in terms of the percentage of subjects with a ≥ 4-fold increase in serum total binding antibody to each of the RSV Proteins F, G and N from Day 1 (baseline) to all time points (Day 29 [28 days after the first dose], Day 57 [28 days after the second dose], and Day 181 [six months after the first dose]).
Time Frame: At Day 29, Day 57 and Day 181
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Percentage of subjects
  RSV Protein F, Day 29 | 83 [61.2 to 95.0] | 92 [73.0 to 99.0] | 96 [78.1 to 99.89] | 0 [0.0 to 14.8] | 100 [85.8 to 100.0] | 92 [73.0 to 99.0] | 86 [65.1 to 97.1] | 0 [0.0 to 14.2] | 87 [66.4 to 97.2] | 100 [85.2 to 100.0] | 100 [85.8 to 100.0] | 0 [0.0 to 14.2]
  RSV Protein F, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein F, Day 57 | 86 [65.1 to 97.1] | 92 [73.0 to 99.0] | 95 [77.2 to 99.88] | 0 [0.0 to 14.8] | 100 [85.8 to 100.0] | 92 [73.0 to 99.0] | 86 [65.1 to 97.1] | 0 [0.0 to 14.8] | 87 [66.4 to 97.2] | 100 [84.6 to 100.0] | 100 [85.8 to 100.0] | 0 [0.0 to 14.2]
  RSV Protein F, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein F, Day 181 | 73 [49.8 to 89.3] | 79 [57.8 to 92.9] | 68 [45.1 to 86.1] | 0 [0.0 to 15.4] | 100 [85.2 to 100.0] | 73 [49.8 to 89.3] | 75 [50.9 to 91.3] | 0 [0.0 to 14.8] | 73 [49.8 to 89.3] | 100 [84.6 to 100.0] | 83 [61.2 to 95.0] | 0 [0.0 to 14.2]
  RSV Protein Ga, Day 29 | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2]
  RSV Protein Ga, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Ga, Day 57 | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2]
  RSV Protein Ga, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Ga, Day 181 | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 16.8] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2]
  RSV Protein Gb, Day 29 | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2]
  RSV Protein Gb, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Gb, Day 57 | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2]
  RSV Protein Gb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Gb, Day 181 | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 16.8] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2]
  RSV Protein N, Day 29 | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2]
  RSV Protein N, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein N, Day 57 | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 14.2]
  RSV Protein N, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein N, Day 181 | 0 [0.0 to 15.4] | 0 [0.0 to 14.2] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 16.8] | 0 [0.0 to 14.8] | 0 [0.0 to 15.4] | 0 [0.0 to 15.4] | 0 [0.0 to 14.8] | 0 [0.0 to 14.2]

18. Secondary Outcome: Percentage of Subjects With Serum Total Binding Antibody Titers to Each of the RSV Proteins F, G, and N Greater Than the 3rd Quartile of Serum Total Binding Antibody Titers to RSV Protein F at Day 1
Description: Immunogenicity was measured in terms of the percentage of subjects at Day 29 (28 days after the first dose), Day 57 (28 days after the second dose) and Day 181 (six months after the first dose), with serum total binding antibody titers to each of the RSV proteins F, G, and N greater than the 3rd quartile of serum total binding antibody titers to RSV protein F at Day 1 (baseline).
Time Frame: At Day 29, Day 57 and Day 181
Population: as for outcome 15
Measure: Number (95% Confidence Interval); unit: Percentage of subjects
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Percentage of subjects
  RSV Protein F, Day 29 | 96 [78.1 to 99.89] | 100 [85.8 to 100.0] | 100 [85.2 to 100.0] | 22 [7.5 to 43.7] | 100 [85.8 to 100.0] | 100 [85.8 to 100.0] | 100 [84.6 to 100.0] | 21 [7.1 to 42.2] | 100 [85.2 to 100.0] | 100 [85.2 to 100.0] | 100 [85.8 to 100.0] | 29 [12.6 to 51.1]
  RSV Protein F, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein F, Day 57 | 95 [77.2 to 99.88] | 100 [85.8 to 100.0] | 100 [84.6 to 100.0] | 30 [13.2 to 52.9] | 100 [85.8 to 100.0] | 100 [85.8 to 100.0] | 100 [84.6 to 100.0] | 13 [2.8 to 33.6] | 100 [85.2 to 100.0] | 100 [84.6 to 100.0] | 100 [85.8 to 100.0] | 25 [9.8 to 46.7]
  RSV Protein F, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein F, Day 181 | 91 [70.8 to 98.9] | 100 [85.8 to 100.0] | 95 [77.2 to 99.88] | 23 [7.8 to 45.4] | 100 [85.2 to 100.0] | 100 [84.6 to 100.0] | 100 [83.2 to 100.0] | 17 [5.0 to 38.8] | 100 [84.6 to 100.0] | 100 [84.6 to 100.0] | 100 [85.2 to 100.0] | 21 [7.1 to 42.2]
  RSV Protein Ga, Day 29 | 30 [13.2 to 52.9] | 38 [18.8 to 59.4] | 22 [7.5 to 43.7] | 22 [7.5 to 43.7] | 25 [9.8 to 46.7] | 21 [7.1 to 42.2] | 14 [2.9 to 34.9] | 29 [12.6 to 51.1] | 35 [16.4 to 57.3] | 13 [2.8 to 33.6] | 29 [12.6 to 51.1] | 38 [18.8 to 59.4]
  RSV Protein Ga, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Ga, Day 57 | 27 [10.7 to 50.2] | 38 [18.8 to 59.4] | 23 [7.8 to 45.4] | 22 [7.5 to 43.7] | 25 [9.8 to 46.7] | 17 [4.7 to 37.4] | 14 [2.9 to 34.9] | 22 [7.5 to 43.7] | 39 [19.7 to 61.5] | 14 [2.9 to 34.9] | 25 [9.8 to 46.7] | 38 [18.8 to 59.4]
  RSV Protein Ga, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Ga, Day 181 | 45 [24.4 to 67.8] | 38 [18.8 to 59.4] | 23 [7.8 to 45.4] | 18 [5.2 to 40.3] | 22 [7.5 to 43.7] | 23 [7.8 to 45.4] | 30 [11.9 to 54.3] | 22 [7.5 to 43.7] | 18 [5.2 to 40.3] | 18 [5.2 to 40.3] | 30 [13.2 to 52.9] | 21 [7.1 to 42.2]
  RSV Protein Gb, Day 29 | 30 [13.2 to 52.9] | 21 [7.1 to 42.2] | 30 [13.2 to 52.9] | 26 [10.2 to 48.4] | 21 [7.1 to 42.2] | 17 [4.7 to 37.4] | 23 [7.8 to 45.4] | 38 [18.8 to 59.4] | 30 [13.2 to 52.9] | 17 [5.0 to 38.8] | 42 [22.1 to 63.4] | 25 [9.8 to 46.7]
  RSV Protein Gb, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Gb, Day 57 | 36 [17.2 to 59.3] | 17 [4.7 to 37.4] | 27 [10.7 to 50.2] | 39 [19.7 to 61.5] | 21 [7.1 to 42.2] | 17 [4.7 to 37.4] | 27 [10.7 to 50.2] | 22 [7.5 to 43.7] | 35 [16.4 to 57.3] | 23 [7.8 to 45.4] | 21 [7.1 to 42.2] | 25 [9.8 to 46.7]
  RSV Protein Gb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Gb, Day 181 | 32 [13.9 to 54.9] | 17 [4.7 to 37.4] | 23 [7.8 to 45.4] | 18 [5.2 to 40.3] | 30 [13.2 to 52.9] | 27 [10.7 to 50.2] | 20 [5.7 to 43.7] | 22 [7.5 to 43.7] | 27 [10.7 to 50.2] | 18 [5.2 to 40.3] | 30 [13.2 to 52.9] | 21 [7.1 to 42.2]
  RSV Protein N, Day 29 | 39 [19.7 to 61.5] | 25 [9.8 to 46.7] | 35 [16.4 to 57.3] | 9 [1.1 to 28.0] | 21 [7.1 to 42.2] | 25 [9.8 to 46.7] | 23 [7.8 to 45.4] | 25 [9.8 to 46.7] | 26 [10.2 to 48.4] | 17 [5.0 to 38.8] | 29 [12.6 to 51.1] | 33 [15.6 to 55.3]
  RSV Protein N, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein N, Day 57 | 45 [24.4 to 67.8] | 33 [15.6 to 55.3] | 50 [28.2 to 71.8] | 17 [5.0 to 38.8] | 8 [1.0 to 27.0] | 25 [9.8 to 46.7] | 27 [10.7 to 50.2] | 9 [1.1 to 28.0] | 22 [7.5 to 43.7] | 14 [2.9 to 34.9] | 21 [7.1 to 42.2] | 17 [4.7 to 37.4]
  RSV Protein N, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein N, Day 181 | 32 [13.9 to 54.9] | 25 [9.8 to 46.7] | 32 [13.9 to 54.9] | 5 [0.12 to 22.8] | 13 [2.8 to 33.6] | 36 [17.2 to 59.3] | 30 [11.9 to 54.3] | 22 [7.5 to 43.7] | 23 [7.8 to 45.4] | 9 [1.1 to 29.2] | 26 [10.2 to 48.4] | 17 [4.7 to 37.4]

19. Secondary Outcome: Ratio of RSV F Serum Nab Titers to Each of the RSV F Serum Total Binding Antibody Titers to RSV Proteins F, G and N
Description: Immunogenicity was measured in terms of the ratio of RSV F serum Nab titers to each of the RSV F serum total binding antibody titers to RSV proteins F, G and N at Days 1, 29, 57 and 181.
Time Frame: At Day 1, Day 29, Day 57 and Day 181
Population: as for outcome 15
Measure: Geometric Mean (95% Confidence Interval); unit: Adjusted Geometric Mean Ratio
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
Number analyzed (Participants) | 23 | 24 | 23 | 23 | 24 | 24 | 22 | 24 | 23 | 23 | 24 | 24
Adjusted Geometric Mean Ratio
  RSV Protein F, Day 1 | 2.79 [2.06 to 3.78] | 3.95 [2.91 to 5.35] | 3.18 [2.33 to 4.34] | 3.32 [2.24 to 4.93] | 2.48 [1.76 to 3.50] | 2.64 [1.87 to 3.71] | 2.83 [1.97 to 4.04] | 3.13 [2.09 to 4.67] | 2.55 [1.93 to 3.39] | 2.00 [1.51 to 2.66] | 2.51 [1.90 to 3.31] | 2.57 [1.90 to 3.47]
  RSV Protein F, Day 29 | 10 [8.42 to 12] | 12 [10 to 15] | 12 [10 to 15] | 2.86 [1.96 to 4.18] | 12 [10 to 13] | 10 [8.97 to 12] | 11 [10 to 13] | 2.82 [1.88 to 4.23] | 9.83 [8.58 to 11] | 9.21 [8.06 to 11] | 9.56 [8.39 to 11] | 2.98 [2.26 to 3.92]
  RSV Protein F, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein F, Day 57 | 8.95 [7.37 to 11] | 11 [9.47 to 14] | 12 [9.58 to 14] | 3.24 [2.13 to 4.95] | 13 [12 to 16] | 13 [11 to 15] | 13 [12 to 16] | 2.61 [1.73 to 3.94] | 11 [9.38 to 12] | 11 [10 to 13] | 11 [9.36 to 12] | 3.11 [2.25 to 4.31]
  RSV Protein F, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein F, Day 181 | 8.37 [6.66 to 11] | 13 [10 to 16] | 11 [8.41 to 13] | 2.96 [1.98 to 4.40] | 10 [8.44 to 12] | 9.76 [8.05 to 12] | 9.91 [8.08 to 12] | 2.93 [2.03 to 4.24] | 8.78 [7.09 to 11] | 11 [8.69 to 13] | 9.58 [7.77 to 12] | 3.36 [2.46 to 4.58]
  RSV Protein Ga, Day 1 | 0.27 [0.19 to 0.38] | 0.27 [0.19 to 0.39] | 0.20 [0.14 to 0.29] | 0.21 [0.12 to 0.35] | 0.19 [0.13 to 0.28] | 0.20 [0.14 to 0.29] | 0.18 [0.12 to 0.27] | 0.25 [0.17 to 0.35] | 0.16 [0.11 to 0.23] | 0.15 [0.10 to 0.21] | 0.18 [0.13 to 0.26] | 0.17 [0.10 to 0.28]
  RSV Protein Ga, Day 29 | 0.073 [0.049 to 0.11] | 0.056 [0.038 to 0.083] | 0.061 [0.040 to 0.091] | 0.18 [0.11 to 0.31] | 0.047 [0.032 to 0.068] | 0.045 [0.031 to 0.067] | 0.039 [0.026 to 0.058] | 0.21 [0.14 to 0.30] | 0.043 [0.029 to 0.064] | 0.029 [0.020 to 0.043] | 0.045 [0.031 to 0.065] | 0.19 [0.12 to 0.31]
  RSV Protein Ga, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Ga, Day 57 | 0.076 [0.049 to 0.12] | 0.057 [0.038 to 0.087] | 0.063 [0.040 to 0.097] | 0.18 [0.11 to 0.31] | 0.059 [0.040 to 0.087] | 0.058 [0.039 to 0.085] | 0.049 [0.033 to 0.073] | 0.18 [0.13 to 0.26] | 0.056 [0.039 to 0.081] | 0.034 [0.023 to 0.049] | 0.047 [0.033 to 0.067] | 0.20 [0.12 to 0.35]
  RSV Protein Ga, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Ga, Day 181 | 0.12 [0.078 to 0.18] | 0.095 [0.064 to 0.14] | 0.11 [0.075 to 0.17] | 0.17 [0.10 to 0.29] | 0.076 [0.052 to 0.11] | 0.097 [0.066 to 0.14] | 0.065 [0.043 to 0.098] | 0.23 [0.17 to 0.32] | 0.074 [0.050 to 0.11] | 0.054 [0.036 to 0.080] | 0.078 [0.053 to 0.12] | 0.20 [0.12 to 0.32]
  RSV Protein Gb, Day 1 | 0.45 [0.31 to 0.67] | 0.48 [0.33 to 0.71] | 0.43 [0.29 to 0.64] | 0.46 [0.30 to 0.71] | 0.38 [0.26 to 0.57] | 0.35 [0.24 to 0.52] | 0.46 [0.30 to 0.69] | 0.43 [0.29 to 0.65] | 0.30 [0.20 to 0.46] | 0.26 [0.17 to 0.40] | 0.31 [0.21 to 0.47] | 0.27 [0.16 to 0.45]
  RSV Protein Gb, Day 29 | 0.13 [0.087 to 0.19] | 0.099 [0.067 to 0.15] | 0.12 [0.082 to 0.18] | 0.43 [0.27 to 0.69] | 0.086 [0.059 to 0.12] | 0.076 [0.053 to 0.11] | 0.090 [0.061 to 0.13] | 0.37 [0.25 to 0.56] | 0.079 [0.051 to 0.12] | 0.061 [0.039 to 0.094] | 0.083 [0.054 to 0.13] | 0.32 [0.19 to 0.53]
  RSV Protein Gb, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein Gb, Day 57 | 0.14 [0.089 to 0.22] | 0.11 [0.069 to 0.16] | 0.13 [0.082 to 0.20] | 0.47 [0.29 to 0.76] | 0.11 [0.074 to 0.16] | 0.098 [0.067 to 0.14] | 0.12 [0.080 to 0.18] | 0.31 [0.20 to 0.48] | 0.10 [0.067 to 0.16] | 0.068 [0.044 to 0.10] | 0.081 [0.054 to 0.12] | 0.34 [0.20 to 0.57]
  RSV Protein Gb, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein Gb, Day 181 | 0.19 [0.12 to 0.29] | 0.17 [0.11 to 0.25] | 0.21 [0.14 to 0.32] | 0.42 [0.26 to 0.67] | 0.16 [0.11 to 0.23] | 0.17 [0.12 to 0.25] | 0.15 [0.10 to 0.23] | 0.39 [0.28 to 0.55] | 0.15 [0.098 to 0.23] | 0.11 [0.072 to 0.17] | 0.14 [0.090 to 0.21] | 0.35 [0.21 to 0.59]
  RSV Protein N, Day 1 | 1.99 [1.44 to 2.74] | 2.40 [1.75 to 3.31] | 2.10 [1.52 to 2.92] | 2.07 [1.33 to 3.22] | 1.51 [1.11 to 2.04] | 1.76 [1.30 to 2.38] | 1.88 [1.37 to 2.58] | 1.82 [1.20 to 2.77] | 1.34 [1.04 to 1.71] | 1.21 [0.94 to 1.56] | 1.59 [1.24 to 2.03] | 1.34 [0.96 to 1.88]
  RSV Protein N, Day 29 | 0.59 [0.42 to 0.82] | 0.47 [0.34 to 0.65] | 0.52 [0.38 to 0.73] | 1.77 [1.12 to 2.79] | 0.36 [0.27 to 0.50] | 0.44 [0.32 to 0.60] | 0.44 [0.32 to 0.60] | 1.70 [1.15 to 2.52] | 0.36 [0.27 to 0.48] | 0.26 [0.20 to 0.35] | 0.39 [0.30 to 0.51] | 1.60 [1.15 to 2.22]
  RSV Protein N, Day 57: number analyzed (Participants) | 22 | 24 | 22 | 23 | 24 | 24 | 22 | 23 | 23 | 22 | 24 | 24
  RSV Protein N, Day 57 | 0.62 [0.43 to 0.89] | 0.53 [0.37 to 0.75] | 0.63 [0.44 to 0.90] | 1.96 [1.23 to 3.11] | 0.43 [0.32 to 0.57] | 0.53 [0.39 to 0.71] | 0.51 [0.37 to 0.70] | 1.36 [0.95 to 1.96] | 0.46 [0.36 to 0.60] | 0.33 [0.26 to 0.43] | 0.43 [0.33 to 0.55] | 1.65 [1.12 to 2.41]
  RSV Protein N, Day 181: number analyzed (Participants) | 22 | 24 | 22 | 22 | 23 | 22 | 20 | 23 | 22 | 22 | 23 | 24
  RSV Protein N, Day 181 | 0.87 [0.61 to 1.24] | 0.73 [0.52 to 1.02] | 0.89 [0.62 to 1.26] | 1.80 [1.13 to 2.88] | 0.54 [0.39 to 0.74] | 0.81 [0.58 to 1.12] | 0.73 [0.52 to 1.03] | 1.75 [1.20 to 2.54] | 0.65 [0.51 to 0.84] | 0.54 [0.42 to 0.70] | 0.69 [0.54 to 0.89] | 1.77 [1.25 to 2.52]

ADVERSE EVENTS:
Time Frame: Solicited local and systemic symptoms: from Day 1 (6 hours) through Day 7 after each vaccination; Unsolicited AEs: from Day 1 through Day 28 after each vaccination; SAEs: from study start (Day 1) to study completion (Day 394).
Arm/Group | RSV F 45 No Adj Group | RSV F 45 Alum Adj Group | RSV F 45 MF59 Adj Group | Placebo 1 Group | RSV F 90 No Adj Group | RSV F 90 Alum Adj Group | RSV F 90 MF59 Adj Group | Placebo 2 Group | RSV F 135 No Adj Group | RSV F 135 Alum Adj Group | RSV F 135 MF59 Adj Group | Placebo 3 Group
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 1/24 | 1/24 | 1/24 | 0/24 | 1/24 | 0/24 | 4/24 | 0/24 | 1/24 | 2/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 23/24 | 24/24 | 24/24 | 23/24 | 24/24 | 24/24 | 24/24 | 21/24 | 23/24 | 24/24 | 23/24 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV F 45 No Adj Group (N=24) | RSV F 45 Alum Adj Group (N=24) | RSV F 45 MF59 Adj Group (N=24) | Placebo 1 Group (N=24) | RSV F 90 No Adj Group (N=24) | RSV F 90 Alum Adj Group (N=24) | RSV F 90 MF59 Adj Group (N=24) | Placebo 2 Group (N=24) | RSV F 135 No Adj Group (N=24) | RSV F 135 Alum Adj Group (N=24) | RSV F 135 MF59 Adj Group (N=24) | Placebo 3 Group (N=24)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cartilage injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Basedow's disease (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic shock (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV F 45 No Adj Group (N=24) | RSV F 45 Alum Adj Group (N=24) | RSV F 45 MF59 Adj Group (N=24) | Placebo 1 Group (N=24) | RSV F 90 No Adj Group (N=24) | RSV F 90 Alum Adj Group (N=24) | RSV F 90 MF59 Adj Group (N=24) | Placebo 2 Group (N=24) | RSV F 135 No Adj Group (N=24) | RSV F 135 Alum Adj Group (N=24) | RSV F 135 MF59 Adj Group (N=24) | Placebo 3 Group (N=24)
Lymphadenopathy (Blood and lymphatic system disorders) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (9) | 1 (1) | 1 (1) | 8 (9) | 5 (7) | 2 (4) | 3 (3) | 4 (7) | 1 (1) | 6 (8) | 5 (9) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (6) | 3 (4) | 5 (5) | 5 (7) | 7 (8) | 7 (9) | 5 (6) | 9 (13) | 7 (8) | 5 (8) | 7 (9) | 5 (7)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Gastrointestinal disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 18 (27) | 21 (32) | 19 (32) | 8 (9) | 17 (27) | 21 (32) | 22 (36) | 5 (5) | 20 (30) | 23 (33) | 19 (32) | 8 (12)
Fatigue (General disorders) | 9 (13) | 10 (14) | 13 (20) | 13 (24) | 10 (23) | 14 (16) | 12 (16) | 11 (22) | 9 (13) | 7 (16) | 12 (21) | 9 (16)
Injection site induration (General disorders) | 8 (9) | 6 (7) | 7 (8) | 1 (2) | 6 (7) | 9 (10) | 6 (8) | 0 (0) | 8 (9) | 9 (13) | 7 (11) | 3 (4)
Injection site erythema (General disorders) | 8 (10) | 5 (6) | 4 (4) | 3 (4) | 5 (5) | 5 (10) | 5 (8) | 2 (2) | 4 (6) | 8 (11) | 4 (5) | 5 (7)
Injection site swelling (General disorders) | 4 (4) | 3 (3) | 3 (5) | 1 (2) | 2 (2) | 2 (3) | 6 (7) | 0 (0) | 8 (11) | 3 (4) | 3 (4) | 2 (2)
Chills (General disorders) | 3 (4) | 1 (1) | 6 (6) | 2 (2) | 3 (3) | 4 (5) | 2 (2) | 1 (3) | 3 (6) | 4 (4) | 5 (5) | 3 (3)
Influenza like illness (General disorders) | 2 (2) | 1 (1) | 6 (7) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 4 (4) | 1 (1) | 3 (3)
Injection site haemorrhage (General disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (2) | 1 (1) | 2 (2) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Malaise (General disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hangover (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 11 (16) | 12 (14) | 10 (11) | 11 (15) | 10 (19) | 13 (15) | 9 (12) | 9 (13) | 9 (10) | 10 (11) | 5 (8) | 9 (12)
Rhinitis (Infections and infestations) | 3 (3) | 4 (5) | 3 (3) | 7 (8) | 7 (10) | 7 (7) | 3 (4) | 12 (14) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
Cystitis (Infections and infestations) | 2 (2) | 2 (5) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (2)
Gastroenteritis (Infections and infestations) | 1 (1) | 3 (3) | 5 (5) | 5 (6) | 3 (3) | 3 (3) | 3 (3) | 5 (6) | 4 (5) | 3 (3) | 4 (4) | 4 (4)
Pharyngitis (Infections and infestations) | 1 (2) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0) | 4 (4) | 4 (4) | 4 (4) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 3 (6) | 4 (6) | 3 (3)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 5 (7) | 6 (6) | 3 (3) | 5 (6) | 4 (4) | 2 (3) | 4 (5) | 5 (6) | 5 (8) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 11 (14) | 11 (26) | 9 (10) | 14 (23) | 14 (31) | 11 (21) | 11 (23) | 12 (24) | 11 (19) | 11 (21) | 13 (21) | 10 (13)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 12 (25) | 11 (31) | 12 (24) | 11 (21) | 11 (14) | 9 (15) | 8 (13) | 11 (14) | 9 (12) | 10 (21) | 12 (22) | 11 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (15) | 6 (10) | 9 (15) | 8 (10) | 8 (10) | 8 (11) | 5 (6) | 2 (3) | 5 (7) | 9 (17) | 7 (14) | 10 (12)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (6) | 5 (5) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 5 (6) | 1 (2) | 4 (6) | 6 (7) | 5 (7)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 1 (1) | 1 (2) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 1 (2) | 2 (2) | 1 (2) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (4) | 1 (1)
Tension headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/79/NCT02298179/Prot_000.pdf
  • Statistical Analysis Plan (2017-10-18): https://cdn.clinicaltrials.gov/large-docs/79/NCT02298179/SAP_001.pdf